CLINICAL TRIAL: NCT07176897
Title: Refractive Accuracy of Toric Intraocular Lens Implantation Using Digital Marking Compared to Conventional Marking
Status: Completed | Type: Observational
Sponsor: Colvard Kandavel Eye Center (Other)
Responsible Party: Principal Investigator, Ganesha Kandavel, Primary Investigator, Colvard Kandavel Eye Center
Other Study IDs: 9216252
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cataract; Astigmatism
Keywords: Cataract; Toric; Astigmatism; Digital Marking; Laser cataract surgery; cataract surgery
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Toric Lens Patients: These patients had selected to have laser cataract surgery with an astigmatism-correcting lens
  Interventions: Diagnostic Test: Normal Toric IOL implantation with digital marking

INTERVENTIONS:
Diagnostic Test: Normal Toric IOL implantation with digital marking — Digital marking was compared to bedside marking, but there was no change in clinical practice. The difference in the marks was measured.

SUMMARY:
To evaluate the postoperative refractive accuracy and intraoperative lens rotational placement of a conventional toric intraoperative marking method compared to digital marking.

DETAILED DESCRIPTION:
Preoperative biometry and planning was assessed with the Argos SS-OCT biometer. The ToriCAM application was also used to mark the patient manually at the bedside. A Mendez marker was used to mark the final axis of the IOL, as calculated by Argos. Digital marking was performed using the VERION image guided system. All subjects received both digital and manual marking, and were implanted with Clareon monofocal toric IOLs (CCWOTx) using the digital marker for final IOL alignment. The primary outcome measure was the difference in degrees between the digital marker and the manual marker as measured intraoperatively. Other outcome measures included IOL rotation, residual astigmatism, absolute prediction error (APE), and monocular visual acuity at 2 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults (50-90 years of age) that were candidates for uncomplicated cataract surgery and planned to be implanted with toric IOLs (CCWOTx, Alcon Vision, LLC)

Exclusion Criteria:

* History of amblyopia
* History of macular disease
* History of glaucoma
* History of corneal disease
* History of prior corneal surgery
* History of diabetes
* History of ocular comorbidity that might hamper post operative visual acuity
* History of previous ocular or refractive surgery with expected post-op VA worse than 0.10 logMAR
* History of irregular corneal astigmatism and keratoconus, or severe/uncontrolled ocular surface disease or dry eye disease.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Los Angeles Ophthalmology General practice all ages > 12 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
difference in degrees between the digital marker and the manual marker as measured intraoperatively | From enrollment to the end of post-operative period at 2 months

SECONDARY OUTCOMES:
IOL rotation | From enrollment to the end of post-operative period at 2 months
Residual Astigmatism | From enrollment to the end of post-operative period at 2 months
Absolute Prediction Error (APE) | From enrollment to the end of post-operative period at 2 months
Monocular Visual Acuity | From enrollment to the end of post-operative period at 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colvard-Kandavel Eye Center, Encino, California
  - Freedom Vision Surgery Center, Encino, California

IPD SHARING:
Plan to Share IPD: No
This data is not relevant to research outside of the study.

REFERENCES:
- [Background] Webers VSC, Bauer NJC, Visser N, Berendschot TTJM, van den Biggelaar FJHM, Nuijts RMMA. Image-guided system versus manual marking for toric intraocular lens alignment in cataract surgery. J Cataract Refract Surg. 2017 Jun;43(6):781-788. doi: 10.1016/j.jcrs.2017.03.041. PMID 28732612
- [Background] Rozema JJ, Gobin L, Verbruggen K, Tassignon MJ. Changes in rotation after implantation of a bag-in-the-lens intraocular lens. J Cataract Refract Surg. 2009 Aug;35(8):1385-8. doi: 10.1016/j.jcrs.2009.03.037. PMID 19631125
- [Background] Titiyal JS, Kaur M, Jose CP, Falera R, Kinkar A, Bageshwar LM. Comparative evaluation of toric intraocular lens alignment and visual quality with image-guided surgery and conventional three-step manual marking. Clin Ophthalmol. 2018 Apr 24;12:747-753. doi: 10.2147/OPTH.S164175. eCollection 2018. PMID 29731603
- [Background] Mayer WJ, Kreutzer T, Dirisamer M, Kern C, Kortuem K, Vounotrypidis E, Priglinger S, Kook D. Comparison of visual outcomes, alignment accuracy, and surgical time between 2 methods of corneal marking for toric intraocular lens implantation. J Cataract Refract Surg. 2017 Oct;43(10):1281-1286. doi: 10.1016/j.jcrs.2017.07.030. Epub 2017 Oct 19. PMID 29056301
- [Background] Kim EC, Hwang KY, Lim SA, Yi R, Joo CK. Accuracy of toric intraocular lens implantation using automated vs manual marking. BMC Ophthalmol. 2019 Aug 3;19(1):169. doi: 10.1186/s12886-019-1175-1. PMID 31376834
- [Background] Ding N, Wang X, Song X. Digital versus slit-beam marking for toric intraocular lenses in cataract surgery. BMC Ophthalmol. 2022 Jul 27;22(1):323. doi: 10.1186/s12886-022-02548-y. PMID 35897093
- [Background] Barbera-Loustaunau E, Basanta I, Vazquez J, Duran P, Costa M, Counago F, Garzon N, Angel Sanchez-Tena M. Time-efficiency assessment of guided toric intraocular lens cataract surgery: pilot study. J Cataract Refract Surg. 2021 Dec 1;47(12):1535-1541. doi: 10.1097/j.jcrs.0000000000000688. PMID 34074992
- [Background] Lehmann RP, Houtman DM. Visual performance in cataract patients with low levels of postoperative astigmatism: full correction versus spherical equivalent correction. Clin Ophthalmol. 2012;6:333-8. doi: 10.2147/OPTH.S28241. Epub 2012 Mar 2. PMID 22399846
- [Background] Kodavoor SK, Divya J, Dandapani R, Ramamurthy C, Ramamurthy S, Sachdev G. Randomized trial comparing visual outcomes of toric intraocular lens implantation using manual and digital marker. Indian J Ophthalmol. 2020 Dec;68(12):3020-3024. doi: 10.4103/ijo.IJO_465_20. PMID 33229690
- [Background] Elhofi AH, Helaly HA. Comparison Between Digital and Manual Marking for Toric Intraocular Lenses: A Randomized Trial. Medicine (Baltimore). 2015 Sep;94(38):e1618. doi: 10.1097/MD.0000000000001618. PMID 26402830
- [Background] Shin DE, Lee JM, Kim TI, Seo KY, Koh K. Efficacy of the Image-Guided Alignment System for a Four-Haptic Hydrophobic Monofocal Toric Intraocular Lens. Eye Contact Lens. 2022 Sep 1;48(9):396-402. doi: 10.1097/ICL.0000000000000901. Epub 2022 May 17. PMID 35580544
- [Background] Terauchi R, Horiguchi H, Ogawa T, Shiba T, Tsuneoka H, Nakano T. Posture-related ocular cyclotorsion during cataract surgery with an ocular registration system. Sci Rep. 2020 Feb 7;10(1):2136. doi: 10.1038/s41598-020-59118-9. PMID 32034232
- [Background] Ma JJ, Tseng SS. Simple method for accurate alignment in toric phakic and aphakic intraocular lens implantation. J Cataract Refract Surg. 2008 Oct;34(10):1631-6. doi: 10.1016/j.jcrs.2008.04.041. PMID 18812110
- [Background] Mozayan E, Lee JK. Update on astigmatism management. Curr Opin Ophthalmol. 2014 Jul;25(4):286-90. doi: 10.1097/ICU.0000000000000068. PMID 24837578
- [Background] Nubile M, Carpineto P, Lanzini M, Calienno R, Agnifili L, Ciancaglini M, Mastropasqua L. Femtosecond laser arcuate keratotomy for the correction of high astigmatism after keratoplasty. Ophthalmology. 2009 Jun;116(6):1083-92. doi: 10.1016/j.ophtha.2009.01.013. Epub 2009 Apr 23. PMID 19395035
- [Background] Budak K, Friedman NJ, Koch DD. Limbal relaxing incisions with cataract surgery. J Cataract Refract Surg. 1998 Apr;24(4):503-8. doi: 10.1016/s0886-3350(98)80292-7. PMID 9584246
- [Background] Schallhorn SC, Hettinger KA, Pelouskova M, Teenan D, Venter JA, Hannan SJ, Schallhorn JM. Effect of residual astigmatism on uncorrected visual acuity and patient satisfaction in pseudophakic patients. J Cataract Refract Surg. 2021 Aug 1;47(8):991-998. doi: 10.1097/j.jcrs.0000000000000560. PMID 34290195

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT07176897/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT07176897/ICF_001.pdf